CLINICAL TRIAL: NCT03693755
Title: Dislocation Rates of Femoral Catheter Placed Sonographically Either In-plane or Out-of-plane: A Prospective Randomized Study
Brief Title: Dislocation Rates of Femoral Catheter Placed Sonographically Either In-plane or Out-of-plane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Aguirre (Other)
Responsible Party: Sponsor-Investigator, Jose Aguirre, PD Dr. med José A. Aguirre, MSc, Senior Consultant Anesthetist, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-00940
Record Dates: First submitted 2018-06-27; First posted 2018-10-03 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Catheter Complications

STUDY DESIGN:
Intervention Model Description: 1 Group will be compared to another
Who Masked: Participant
Masking Description: The Patient will not be told in which Group he belongs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-plane Group (Active Comparator): In this Group the femoral nerve catheter will be placed with the in-plane technique.
  Interventions: Procedure: In-plane Group; Procedure: Out-of-plane Group
- Out-of-plane Group (Active Comparator): In this Group the femoral nerve catheter will be placed with the out-of-plane technique.
  Interventions: Procedure: In-plane Group; Procedure: Out-of-plane Group

INTERVENTIONS:
Procedure: In-plane Group — Placement of femoral nerve catheter under ultrasound control
Procedure: Out-of-plane Group — Placement of femoral nerve catheter under ultrasound control

SUMMARY:
Dislocation of the femoral nerve catheters, which are used as postoperative analgesic method after knie surgery, will be studied. Two Groups will be compared; in the first group the femoral nerve catheter will be placed sonographically with the in-plane technique, whereas in the other Group the femoral nerve catheter will be placed sonographically with the out-of-plane technique

DETAILED DESCRIPTION:
Patients scheduled for elective major knee surgery will be assessed for eligibility and after written informed consent included in this clinical trial. Prior to surgery, the patient will receive a femoral catheter with either ultrasound placed in-plane (IP) or with ultrasound placed out-of-plane (OOP) as perioperative analgesic regimen using well-established and previously published techniques. The allocation to the different groups will be according to a computerized random-list established the day prior to surgery. In all cases, continuous regional anaesthesia regimen will be started after surgery. For surgery the patient can receive spinal anaesthesia, or a general anaesthesia. The use of a sciatic block will be applied according to the clinical standards of our department. Ropivacaine 0.3% (bag with 100 ml, Sintetica SA, Mendrisio Switzerland) 20 ml for the femoral catheter insertion. In both groups 10ml of ropivacaine 0.3% will be applied over the needle and 10ml over the catheter after its placement. In both groups the catheters will be connected to the electronic pump in the recovery room and run with ropivacaine 0.3% at 6 ml/h with boli of 4ml every 20min.

First rescue medication: ropivacaine 0.3% 20ml up to 3 x day. The catheters will stay in place for 48 hours and removed only if VAS< 40 with standard analgesia.

At 24 and 48 hours after placement of the femoral catheter, a bolus of NaCl 0.9% 10ml will be applied under ultrasound control in both groups and dislocation will be noted if the local anaesthetic does not reach the femoral nerve. In that case it will be noted where the local anaesthetic is localised. Block quality will be checked by applying cold on the front of the knee and measuring the sensation to cold in a scale from 0 to 2 (before NaCl 0.9% application). Pain will be assessed before the dislocation test only for in front and medial side of the knee in a regularly used NRS scale from 0 to 10. Complications and side effects of regional anesthesia in both groups will be documented (toxicity, blood in catheter, infection).

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists class I-III patients, both sexes

≥ 18 years old

* Patients are undergoing major knie surgery at our University Hospital with standard use of regional anesthesia techniques to provide analgesia

Exclusion Criteria:

* Contraindications or allergy to the use of local anesthetics or other drugs used in the study.
* Women who are pregnant or breast feeding
* Women who have the intention to become pregnant during the course of the study
* Lack of safe contraception, defined as: female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator(s) in individual cases
* Patients with acute porphyria
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrollment into the current study
* BMI > 40
* Local inflammation in the inguinal area
* Patient refusal for regional anesthesia or participation in the study
* Enrollment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Dislocation of the femoral nerve catheter at 48 hours after its placement. | 48 hours after the placement of the catheter
  The catheter will be checked if in the right place using ultrasound location

SECONDARY OUTCOMES:
Time to place the catheter | 30min (time needed to place and fix a femoral catheter)
  Time to place the catheter measured in seconds
satisfaction of the patient | 48 hours after the placement of the catheter
  satisfaction of the Patient during the block procedure in a scale of 0 to 10 (0 being not satisfied at all and 10 being totally satisfied)
number of failed blocks | 30min (time needed to place and fix a femoral catheter and regognize if it works)
  number of failed blocks needed to be repeated
difficulty placing the catheter | 30min (time needed to place and fix a femoral catheter and to decide if it was difficult)
  difficulty placing the catheter under ultrasound control
Effect of the femoral catheter on the sensory sensation | at 24 hours and 48 hours after the femoral nerve catheter
  cold (cold metal bar) and pinprick (atraumatic test, using a sharp tip): can the patient recognize cold and sharp during the femoral nerve block? Answers are yes or no.
rescue boli given over the catheter in the 48 hours after its placement | At 48 hours after the placement of the catheter
  amount of local anaesthetic rescue boli given
Dislocation of the femoral nerve catheter at 24 hours after its placement. | At 24 and at 48 hours after the placement of the catheter
  amount of catheter dislocations

CONTACTS AND LOCATIONS:
Overall Officials: Urs Eichenberger, Prof. Dr. med., Study Chair — Department of Anaesthesia, Intensive Care and Pain Medicine
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalimeris K, Rupnik B, Allenspach K, Fucentese SF, Gotschi T, Aguirre J, Eichenberger U. Dislocation rates of perineural catheters placed either perpendicular or parallel to the femoral nerve: A randomised controlled trial. Eur J Anaesthesiol. 2020 Sep;37(9):758-764. doi: 10.1097/EJA.0000000000001237. PMID 32453168